CLINICAL TRIAL: NCT01339910
Title: A Randomized, Multi-Center, Phase III Study of Allogeneic Stem Cell Transplantation Comparing Regimen Intensity in Patients With Myelodysplastic Syndrome or Acute Myeloid Leukemia (BMT CTN #0901)
Brief Title: Reduced Intensity Regimen vs Myeloablative Regimen for Myeloid Leukemia or Myelodysplastic Syndrome (BMT CTN 0901)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Accrual terminated as recommended by the data and safety monitoring board.
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Cancer Institute (NCI) (NIH); Blood and Marrow Transplant Clinical Trials Network (Network); National Marrow Donor Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMTCTN0901; U01HL069294 (NIH); U01HL069294-05 (NIH); BMT CTN 0901 (Other: Blood and Marrow Transplant Clinical Trial Network); 5U24CA076518 (NIH)
Record Dates: First submitted 2011-04-20; First posted 2011-04-21 (Estimated); Results first posted 2018-05-30 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2022-12

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Acute Myelogenous Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — fludarabine; Busulfan; fludarabine phosphate; Melphalan; Cyclophosphamide; Whole-Body Irradiation; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Reduced Intensity Conditioning (RIC) (Experimental): One of two different regimens in RIC will be administered; fludarabine and busulfan, or fludarabine and melphalan.
  Interventions: Drug: Fludarabine and Busulfan; Drug: Fludarabine and Melphalan
- Myeloablative Conditioning Regimen (MAC) (Active Comparator): One of three different regimens in MAC will be administered; busulfan and fludarabine, busulfan and cyclophosphamide, or cyclophosphamide and total body irradiation.
  Interventions: Drug: Busulfan and Fludarabine; Drug: Busulfan and Cyclophosphamide; Drug: Cyclophosphamide and Total Body Irradiation

INTERVENTIONS:
Drug: Fludarabine and Busulfan — (Flu/Bu)
  * Fludarabine: 30 mg/m^2/day on Days -6 to -2 (total dose of 150 mg/m^2)
  * Busulfan: 4 mg/kg/day PO or 3.2 mg/kg/day (total dose of 8 mg/kg or 6.4 mg/kg, respectively) on Days -5 to -4
  Other Names: Fludara and Busulfex
  Arms: Reduced Intensity Conditioning (RIC)
Drug: Fludarabine and Melphalan — (Flu/Mel)
  * Fludarabine: 30 mg/m^2/day on Days -5 to -2 (total dose of 120 mg/m^2)
  * Melphalan: 140 mg/m^2 on Day -2
  Other Names: Fludara and Alkeran
  Arms: Reduced Intensity Conditioning (RIC)
Drug: Busulfan and Fludarabine — (Bu/Flu)
  * Busulfan: 4 mg/kg/day PO, 3.2 mg/kg/day IV or mg/m^2/day with Bu Css 900±100 ng/mL (total dose of 16 mg/kg, 12.8 mg/kg or 520 mg/m^2, respectively) on Days -5 to -2
  * Fludarabine: 30 mg/m^2/day on Days -5 to -2: Flu (total dose of 120 mg/m^2)
  Other Names: Busulfex and Fludara
  Arms: Myeloablative Conditioning Regimen (MAC)
Drug: Busulfan and Cyclophosphamide — (Bu/Cy)
  * Busulfan: 4 mg/kg/day PO, 3.2 mg/kg/day IV or 130 mg/m^2/day with Bu Css 900 ± 100 ng/mL (total dose of 16 mg/kg or 12.8 mg/kg or 520 mg/m^2, respectively) on Days -7 to -4
  * Cyclophosphamide: 60 mg/kg/day on Days -3 to -2 (total dose of 120 mg/kg)
  Other Names: Busulfex and Cytoxan
  Arms: Myeloablative Conditioning Regimen (MAC)
Drug: Cyclophosphamide and Total Body Irradiation — (Cy/TBI)
  * TBI: 1200-1420 cGy on Days -7 to -4
  * Cyclophosphamide: 60 mg/kg/day on Days -3 to -2 (total dose of 120 mg/kg)
  Other Names: Cytoxan and radiation
  Arms: Myeloablative Conditioning Regimen (MAC)

SUMMARY:
The study is designed as a Phase III, multicenter trial comparing outcomes after allogeneic hematopoietic stem cell transplantation (HCT) for acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS) between patients receiving myeloablative conditioning (MAC) versus reduced intensity conditioning (RIC) regimens.

DETAILED DESCRIPTION:
Patients randomized to RIC will receive one of two regimen types: the combination of fludarabine (120-180 mg/m^2) and busulfan (less than or equal to 8 mg/kg or IV equivalent) (Flu/Bu) or fludarabine (120-180 mg/m^2) and melphalan (less than 150 mg/m^2) (Flu/Mel). Patient randomized to MAC will receive one of three regimens: busulfan (16 mg/kg oral or 12.8 mg/kg IV equivalent) and cyclophosphamide (120 mg/kg) (Bu/Cy); or, busulfan (16 mg/kg PO or 12.8 mg/kg IV) and fludarabine (120-180 mg/m^2) (Bu/Flu); or, cyclophosphamide (120 mg/kg) and total body irradiation (greater than 1200-1420cGy) (CyTBI). A total of 356 patients (178 to each arm) will be accrued on this study over a period of four years. Patients will be followed for up to 18 months from transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or less than 65 years old and equal to or greater than 18 years old.
* Patients with the diagnosis of MDS or AML with fewer than 5% myeloblasts in the bone marrow and no leukemic myeloblasts in the peripheral blood on morphologic analysis performed within 30 days of start of the conditioning regimen enrollment.
* For patients receiving treatment of their MDS or AML prior to transplantation: a)Interval between the start of the most recent cycle of conventional cytotoxic chemotherapy and enrollment must be at least 30 days; b)Interval between completing treatment with a hypomethylating agent or other non-cytotoxic chemotherapy and enrollment must be at least 10 days.
* Patients must have a related or unrelated bone marrow or peripheral blood donor who is human leukocyte antigen (HLA)-matched at 7 or 8 of 8 HLA-A, -B, -C and -DRB1 at high resolution using DNA-based typing.
* HCT-Specific Comorbidity Index Score (HCT-CI) less than or equal to 4.
* Organ function: a) Cardiac function: Ejection fraction greater than or equal to 40%; b) Hepatic function: total bilirubin less than or equal to 2 times the upper limit of normal and alanine aminotransferase (ALT) and aspartate aminotransferase (AST) less than or equal to 3 times the upper limit of normal.; c)Pulmonary function: Diffusing capacity of the lung for carbon monoxide (DLCO) greater than or equal to 40% and forced expiratory volume in one second (FEV1) greater than or equal to 50% (corrected for hemoglobin).
* Creatinine clearance greater than or equal to 50mL/min based on the Cockcroft-Gault formula.
* Signed informed consent.

Exclusion Criteria:

* Prior allograft or prior autograft.
* Symptomatic coronary artery disease.
* Leukemia involvement in the central nervous system (CNS) within 4 weeks of enrollment for patients with a history of prior CNS leukemia involvement (i.e., leukemic blasts previously detected in the cerebral spinal fluid).
* Karnofsky Performance Score less than 70.
* Patients receiving supplemental oxygen.
* Planned use of donor lymphocyte infusion (DLI) therapy.
* Patients with uncontrolled bacterial, viral or fungal infections (undergoing appropriate treatment and with progression of clinical symptoms).
* Patients seropositive for the human immunodeficiency virus (HIV).
* Patients with prior malignancies, except resected basal cell carcinoma or treated cervical carcinoma in situ. Cancer treated with curative intent greater than 5 years previously. Cancer treated with curative intent less than 5 years previously will not be allowed unless approved by the Protocol Officer or one of the Protocol Chairs.
* Females who are pregnant or breastfeeding.
* Fertile men and women unwilling to use contraceptive techniques during and for 12 months following treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2017-01-16 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Horowitz, MD, Study Director — Center for International Blood and Marrow Transplant Research
Locations (32):
- United States (32):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - University of California, San Diego Medical Center, La Jolla, California
  - University of Florida College of Medicine, Gainesville, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Blood and Marrow Transplant Program at Northside Hospital, Atlanta, Georgia
  - University of Kansas, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - DFCI, Brigham & Women's Hospital, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University/Barnes Jewish Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Roswell Park Cancer Institute, Buffalo, New York
  - Mount Sinai Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Hospital at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Jewish Hospital BMT Program, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Utah BMT/University of Utah Medical School, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - University of Wisconsin Hospital & Clinics, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Findings will be published in a manuscript
Time Frame: Within 6 months of official study closure at participating sites.
Access Criteria: Available to the public.
URL: https://biolincc.nhlbi.nih.gov/home/

REFERENCES:
- [Background] Vardiman JW, Thiele J, Arber DA, Brunning RD, Borowitz MJ, Porwit A, Harris NL, Le Beau MM, Hellstrom-Lindberg E, Tefferi A, Bloomfield CD. The 2008 revision of the World Health Organization (WHO) classification of myeloid neoplasms and acute leukemia: rationale and important changes. Blood. 2009 Jul 30;114(5):937-51. doi: 10.1182/blood-2009-03-209262. Epub 2009 Apr 8. PMID 19357394
- [Background] Sorror ML, Maris MB, Storb R, Baron F, Sandmaier BM, Maloney DG, Storer B. Hematopoietic cell transplantation (HCT)-specific comorbidity index: a new tool for risk assessment before allogeneic HCT. Blood. 2005 Oct 15;106(8):2912-9. doi: 10.1182/blood-2005-05-2004. Epub 2005 Jun 30. PMID 15994282
- [Background] Filipovich AH, Weisdorf D, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. Biol Blood Marrow Transplant. 2005 Dec;11(12):945-56. doi: 10.1016/j.bbmt.2005.09.004. PMID 16338616
- [Background] Copelan E, Casper JT, Carter SL, van Burik JA, Hurd D, Mendizabal AM, Wagner JE, Yanovich S, Kernan NA. A scheme for defining cause of death and its application in the T cell depletion trial. Biol Blood Marrow Transplant. 2007 Dec;13(12):1469-76. doi: 10.1016/j.bbmt.2007.08.047. PMID 18022577
- [Result] Scott BL, Pasquini MC, Logan BR, Wu J, Devine SM, Porter DL, Maziarz RT, Warlick ED, Fernandez HF, Alyea EP, Hamadani M, Bashey A, Giralt S, Geller NL, Leifer E, Le-Rademacher J, Mendizabal AM, Horowitz MM, Deeg HJ, Horwitz ME. Myeloablative Versus Reduced-Intensity Hematopoietic Cell Transplantation for Acute Myeloid Leukemia and Myelodysplastic Syndromes. J Clin Oncol. 2017 Apr 10;35(11):1154-1161. doi: 10.1200/JCO.2016.70.7091. Epub 2017 Feb 13. PMID 28380315

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between June 2011 and April 2014 from 32 transplant centers
Groups:
- Myeloablative Conditioning Regimen (MAC): One of three different regimens in MAC will be administered; busulfan and fludarabine, busulfan and cyclophosphamide, or cyclophosphamide and total body irradiation.
  Busulfan and Fludarabine: (Bu/Flu)
  * Busulfan: 4 mg/kg/day PO, 3.2 mg/kg/day IV or mg/m^2/day with Bu Css 900±100 ng/mL (total dose of 16 mg/kg, 12.8 mg/kg or 520 mg/m^2, respectively) on Days -5 to -2
  * Fludarabine: 30 mg/m^2/day on Days -5 to -2: Flu (total dose of 120 mg/m^2)
  Busulfan and Cyclophosphamide: (Bu/Cy)
  * Busulfan: 4 mg/kg/day PO, 3.2 mg/kg/day IV or 130 mg/m^2/day with Bu Css 900 ± 100 ng/mL (total dose of 16 mg/kg or 12.8 mg/kg or 520 mg/m^2, respectively) on Days -7 to -4
  * Cyclophosphamide: 60 mg/kg/day on Days -3 to -2 (total dose of 120 mg/kg)
  Cyclophosphamide and Total Body Irradiation: (Cy/TBI)
  * TBI: 1200-1420 cGy on Days -7 to -4
  * Cyclophosphamide: 60 mg/kg/day on Days -3 to -2 (total dose of 120 mg/kg)
- Reduced Intensity Conditioning (RIC): One of two different regimens in RIC will be administered; fludarabine and busulfan, or fludarabine and melphalan.
  Fludarabine and Busulfan: (Flu/Bu)
  * Fludarabine: 30 mg/m^2/day on Days -6 to -2 (total dose of 150 mg/m^2)
  * Busulfan: 4 mg/kg/day PO or 3.2 mg/kg/day (total dose of 8 mg/kg or 6.4 mg/kg, respectively) on Days -5 to -4
  Fludarabine and Melphalan: (Flu/Mel)
  * Fludarabine: 30 mg/m^2/day on Days -5 to -2 (total dose of 120 mg/m^2)
  * Melphalan: 140 mg/m^2 on Day -2
Period: Overall Study
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Started | 135 | 137
Completed | 132 | 133
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Disease relapse | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC) | Total
Number analyzed (Participants) | 135 | 137 | 272
Age, Continuous [Median (Full Range); unit: years] | 54.8 [21.9 to 66.0] | 54.8 [21.9 to 65.9] | 54.8 [21.9 to 66.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 70 | 129
  Male | 76 | 67 | 143
Primary Disease [Count of Participants; unit: Participants]
  Acute Myeloid Leukemia (AML) | 108 | 110 | 218
  Myelodysplastic Syndrome (MDS) | 27 | 27 | 54
MDS WHO Classification [Count of Participants; unit: Participants] — Participants with MDS are categorized per 2008 WHO classification (Vardiman et al. 2009). Major features of each class are given below:
  Refractory Anemia (RA): Anemia without marrow blasts or sideroblasts; Refractory Anemia with Ringed Sideroblasts (RARS): > 15% marrow sideroblasts; Refractory Cytopenias with Multilineage Dysplasia (RCMD): Dysplasia in >10% marrow cells; Isolated del(5q) (Del-5q): Isolated del(5q) in marrow; Unclassified (MDS-U) Refractory Anemia with Excess Blasts-1 (RAEB-1): 5-9% marrow blasts; Refractory Anemia with Excess Blasts-2 (RAEB-2): 10-19% marrow blasts; Population: Participants with MDS
  Participants
    number analyzed (Participants) | 27 | 27 | 54
    RA/RARS/RCMD/RCMD-RS/Del-5q/MDS-U | 16 | 17 | 33
    RAEB-1 | 5 | 5 | 10
    RAEB-2 | 6 | 5 | 11
AML WHO Classification [Count of Participants; unit: Participants] — Participants with AML are categorized per 2008 WHO classification (Vardiman et al. 2009). Major features of each class are given below:
  AML with recurrent genetic abnormalities: Presence of specific genetic abnormalities known to be prognostic; AML with multilineage dysplasia: > 50% of cells in at least 2 myeloid lineages are dysplastic; AML and MDS, therapy related: development of myeloid neoplasms in response to therapy that is diagnosed as either AML or MDS; AML not otherwise specified: AML that does not satisfy criteria for other classes Population: Participants with AML
  Participants
    number analyzed (Participants) | 108 | 110 | 218
    AML with recurrent genetic abnormalities | 12 | 20 | 32
    AML with multilineage dysplasia | 8 | 12 | 20
    AML and MDS, therapy related | 2 | 3 | 5
    AML, not otherwise specified | 86 | 75 | 161
Disease Duration [Median (Full Range); unit: months] | 6 [2 to 86] | 6 [2 to 130] | 6 [2 to 130]
Disease Risk Status [Count of Participants; unit: Participants] — Disease risk status is defined according to cytogenetic and molecular abnormalities identified prior to transplantation and classified as standard or high risk. Among AML participants, high-risk disease is defined as the presence of cytogenetic abnormalities at 3q, 9q, 11q, 20q, 21q, or 17p; the presence of del(5q)/-5, -7/del(7q), t(6;9), or t(9;22); and/or FLT-3 internal tandem duplication mutation. Among MDS participants, high-risk disease is defined as the presence of > 10% blasts in bone marrow.
  Participants
    Standard | 74 | 71 | 145
    High | 54 | 61 | 115
    Unknown | 7 | 5 | 12
HCT-CI [Count of Participants; unit: Participants] — The Hematopoietic Cell Transplantation-specific Comorbidity Index (HCT-CI) (Sorror et al., 2005) summarizes relevant comorbidities present in participants prior to allogeneic transplant. Each comorbidity reported at the time of transplant is given a score of 0, 1, 2, or 3 and the overall HCT-CI score is the sum of the comorbidity scores, ranging from 0 - 26.
  Participants
    0 | 46 | 40 | 86
    1-2 | 45 | 52 | 97
    3 or more | 42 | 44 | 86
    Unknown | 2 | 1 | 3
Conditioning Regimen [Count of Participants; unit: Participants] — Flu/Bu4: busulfan (16 mg/kg oral or 12.8 mg/kg IV) and fludarabine (120-180 mg/m2); Bu/Cy: busulfan (16 mg/kg oral or 12.8 mg/kg IV) and cyclophosphamide (120 mg/kg) ; Cy/TBI: cyclophosphamide (120 mg/kg) and total body irradiation (1200-1420 cGy); Flu/Mel: fludarabine (120-180 mg/m2) and melphalan (≤ 150 mg/m2); Flu/Bu2: fludarabine (120-180 mg/m2) with busulfan (≤ 8 mg/kg oral or 6.4 mg/kg IV);
  Flu/Bu4, Bu/Cy, and Cy/TBI are myeloablative conditioning regimens, while Flu/Mel and Flu/Bu2 are reduced intensity conditioning regimens.
  Participants
    Flu/Bu4 | 87 | 0 | 87
    Bu/Cy | 40 | 0 | 40
    Cy/TBI | 8 | 0 | 8
    Flu/Mel | 0 | 27 | 27
    Flu/Bu2 | 0 | 110 | 110
GVHD Prophylaxis [Count of Participants; unit: Participants] — Prophylaxis for Graft Versus Host Disease
  Participants
    Tacrolimus / Methotrexate | 110 | 112 | 222
    Cyclosporine / Methotrexate | 3 | 3 | 6
    TAC / Mycophenolate mofetil | 8 | 5 | 13
    Cyclosporine / Mycophenolate mofetil | 1 | 0 | 1
    Sirolimus / Tacrolimus | 10 | 12 | 22
    Other | 3 | 5 | 8
ATG Use [Count of Participants; unit: Participants] — Use of Anti-Thymocyte Globulin
  Participants
    Yes | 18 | 22 | 40
    No | 117 | 115 | 232
Donor Type [Count of Participants; unit: Participants]
  Matched Related | 57 | 58 | 115
  Mismatched Related | 2 | 5 | 7
  Matched Unrelated | 66 | 58 | 124
  Mismatched Unrelated | 10 | 16 | 26
Donor Source [Count of Participants; unit: Participants]
  Peripheral Blood | 127 | 123 | 250
  Bone Marrow | 8 | 14 | 22

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Overall survival is defined as survival of death from any cause.
Time Frame: 18 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 135 | 137
percentage | 77.5 [69.4 to 83.7] | 67.7 [59.1 to 74.9]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in overall survival at 18 months post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. 18 month overall survival was compared between treatment arms using the difference in Kaplan-Meier estimators, which should be close to 0 under the null hypothesis; Test type: Superiority; p = 0.07, Difference in Kaplan-Meier estimators — This final test was performed at a 0.049 significance level, since 0.001 was spent at interim analyses and the overall significance level was 0.050; Difference in 18 month OS (MAC-RIC) = 9.8, 95% CI 2-sided [-0.8 to 20.3]

2. Secondary Outcome: Percentage of Participants With Relapse-Free Survival (RFS)
Description: Relapse-free survival is defined as survival without relapse of the primary disease.
Time Frame: 18 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 135 | 137
percentage | 67.8 [59.1 to 75.0] | 47.3 [38.7 to 55.4]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in relapse-free survival at 18 months post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. 18 month relapse-free survival was compared between treatment arms using the difference in Kaplan-Meier estimators, which should be close to 0 under the null hypothesis; Test type: Superiority; p < 0.01, Difference in Kaplan-Meier estimators — Test performed at a significance level of 0.05; Difference in 18 month RFS (MAC-RIC) = 20.4, 95% CI 2-sided [8.9 to 32.0]

3. Secondary Outcome: Percentage of Participants With Disease Relapse
Description: Disease Relapse is defined as relapse of the primary disease.
Time Frame: 18 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 135 | 137
percentage | 13.5 [8.3 to 19.8] | 48.3 [39.6 to 56.4]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of disease relapse during the first 18 months post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of disease relapse was compared between treatment arms using Gray's test, treating death as a competing risk; Test type: Superiority; p < 0.001, Gray's test — Test performed at a significance level of 0.05

4. Secondary Outcome: Percentage of Participants With Treatment-related Mortality
Description: Treatment-related mortality is defined as death without a previous relapse of the primary disease.
Time Frame: 18 months post-randomization
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 135 | 137
percentage | 15.8 [10.2 to 22.5] | 4.4 [1.8 to 8.9]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of treatment-related mortality during the first 18 months post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of treatment-related mortality was compared between treatment arms using Gray's test, treating disease relapse as a competing risk; Test type: Superiority; p = 0.002, Gray's test — Test performed at a significance level of 0.05

5. Secondary Outcome: Percentage of Participants With Neutrophil and Platelet Engraftment
Description: Neutrophil engraftment is defined as achieving an absolute neutrophil count greater than 500x10^6/liter for 3 consecutive measurements on different days. The first of the 3 days will be designated the day of neutrophil engraftment. Platelet engraftment is defined as achieving platelet counts greater than 20,000/microliter for consecutive measurements over 7 days without requiring platelet transfusions. The first of the 7 days will be designated the day of platelet engraftment. Subjects must not have had platelet transfusions during the preceding 7 days.
Time Frame: Days 28 and 60 post-transplant
Population: Transplanted participants
Measure: Number; unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
percentage
  Neutrophil Engraftment at Day 28 | 98.5 | 97.8
  Platelet Engraftment at Day 60 | 95.5 | 96.2
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of neutrophil engraftment at Day 28 post-transplant between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of neutrophil engraftment at Day 28 was compared between treatment arms using the difference in Aalen-Johansen estimators, which should be close to 0 under the null hypothesis. Death was treated as a competing risk; Test type: Superiority; p = 0.002, Difference in Aalen-Johansen estimators — Test performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of platelet engraftment at Day 60 post-transplant between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of platelet engraftment at Day 60 was compared between treatment arms using the difference in Aalen-Johansen estimators, which should be close to 0 under the null hypothesis. Death was treated as a competing risk; Test type: Superiority; p = 0.065, Difference in Aalen-Johansen estimators — Test performed at a significance level of 0.05

6. Secondary Outcome: Number of Participants With Donor Cell Engraftment
Description: Donor cell engraftment will be assessed by donor-recipient chimerism assays. Full donor chimerism is defined as the presence of at least 95% donor cells as a proportion of the total population in the peripheral blood or bone marrow. Graft rejection is defined as the presence of no more than 5% donor cells as a proportion of the total population. Mixed chimerism is defined as the presence of between 5% and 95% donor cells. Mixed or full donor chimerism will be considered evidence of donor engraftment.
Time Frame: Days 28 and 100 and 18 months post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants
  Day 28: Full Donor Chimerism | 86 | 80
  Day 28: Mixed Chimerism | 9 | 30
  Day 28: Graft Rejection | 1 | 1
  Day 28: Death Prior to Assessment | 0 | 0
  Day 28: Unknown (relapsed or missing assay) | 36 | 22
  Day 100: Full Donor Chimerism | 106 | 86
  Day 100: Mixed Chimerism | 12 | 30
  Day 100: Graft Rejection | 2 | 1
  Day 100: Death Prior to Assessment | 6 | 8
  Day 100: Unknown (relapsed or missing assay) | 6 | 8
  18 Months: Full Donor Chimerism | 71 | 66
  18 Months: Mixed Chimerism | 4 | 5
  18 Months: Graft Rejection | 1 | 1
  18 Months: Death Prior to Assessment | 31 | 42
  18 Months: Unknown (relapsed or missing assay) | 25 | 19
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the proportions of participants with full chimerism, mixed chimerism, graft rejection, and death prior to assessment at Day 28 post-transplant between AML/MDS participants receiving MAC and RIC conditioning regimens; Test type: Superiority; p = 0.005, Chi-squared — Test performed at a significance level of 0.05; 3 degrees of freedom
Statistical Analysis 2: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the proportions of participants with full chimerism, mixed chimerism, graft rejection, and death prior to assessment at Day 100 post-transplant between AML/MDS participants receiving MAC and RIC conditioning regimens; Test type: Superiority; p = 0.011, Chi-squared — Test performed at a significance level of 0.05; 3 degrees of freedom
Statistical Analysis 3: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the proportions of participants with full chimerism, mixed chimerism, graft rejection, and death prior to assessment at 18 months post-transplant between AML/MDS participants receiving MAC and RIC conditioning regimens; Test type: Superiority; p = 0.39, Chi-squared — Test performed at a significance level of 0.05; 3 degrees of freedom

7. Secondary Outcome: Percentage of Participants With Acute Graft Versus Host Disease (GVHD)
Description: Acute GVHD is graded according to the scoring system proposed by Przepiorka et al.1995:
  Skin stage:
  0: No rash
  1. Rash <25% of body surface area
  2. Rash on 25-50% of body surface area
  3. Rash on > 50% of body surface area
  4. Generalized erythroderma with bullous formation
  Liver stage (based on bilirubin level)*:
  0: <2 mg/dL
  1. 2-3 mg/dL
  2. 3.01-6 mg/dL
  3. 6.01-15.0 mg/dL
  4. >15 mg/dL
  GI stage*:
  0: No diarrhea or diarrhea <500 mL/day
  1. Diarrhea 500-999 mL/day or persistent nausea with histologic evidence of GVHD
  2. Diarrhea 1000-1499 mL/day
  3. Diarrhea >1500 mL/day
  4. Severe abdominal pain with or without ileus * If multiple etiologies are listed for liver or GI, the organ system is downstaged by 1.
  GVHD grade:
  0: All organ stages 0 or GVHD not listed as an etiology I: Skin stage 1-2 and liver and GI stage 0 II: Skin stage 3 or liver or GI stage 1 III: Liver stage 2-3 or GI stage 2-4 IV: Skin or liver stage 4
Time Frame: Day 100 post-transplant
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
percentage
  Grade II-IV Acute GVHD | 44.7 [36.0 to 53.0] | 31.6 [23.8 to 39.6]
  Grade III-IV Acute GVHD | 13.6 [8.0 to 20.0] | 6.8 [3.0 to 12.0]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of grade II-IV acute GVHD during the first 100 days post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of grade II-IV acute GVHD was compared between treatment arms using Gray's test, treating death as a competing risk; Test type: Superiority; p = 0.024, Gray's test — Test performed at a significance level of 0.05
Statistical Analysis 2: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of grade III-IV acute GVHD during the first 100 days post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of grade III-IV acute GVHD was compared between treatment arms using Gray's test, treating death as a competing risk; Test type: Superiority; p = 0.066, Gray's test — Test performed at a significance level of 0.05

8. Secondary Outcome: Percentage of Participants With Chronic GVHD
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe. Occurrence of chronic GVHD is defined as the occurrence of mild, moderate, or severe chronic GVHD per this classification.
Time Frame: 18 months post-transplant
Population: Transplanted participants
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
percentage | 64.0 [55.0 to 71.7] | 47.6 [38.8 to 58.8]
Statistical Analysis 1: Comparison: Myeloablative Conditioning Regimen (MAC) vs Reduced Intensity Conditioning (RIC); The null hypothesis is that there is no difference in the cumulative incidence of chronic GVHD during the first 18 months post-randomization between AML/MDS participants receiving MAC and RIC conditioning regimens. Cumulative incidence of chronic GVHD was compared between treatment arms using Gray's test, treating death as a competing risk; Test type: Superiority; p = 0.019, Gray's test — Test performed at a significance level of 0.05

9. Secondary Outcome: Number of Participants With Chronic GVHD Severity
Description: Chronic GVHD is classified per 2005 NIH Consensus Criteria (Filipovich et al. 2005) into categories of severity: none, mild, moderate, and severe.
Time Frame: 18 months post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants
  None | 47 | 70
  Mild | 40 | 34
  Moderate | 33 | 17
  Severe | 12 | 12

10. Secondary Outcome: Number of Participants With Primary Graft Failure
Description: Primary graft failure is defined by lack of neutrophil engraftment.
Time Frame: 28 days post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants | 1 | 3

11. Secondary Outcome: Number of Participants With Secondary Graft Failure
Description: Secondary graft failure is defined by initial neutrophil engraftment followed by subsequent decline in neutrophil counts to less than 500x10^6/liter that is unresponsive to growth factor therapy.
Time Frame: 18 months post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants | 1 | 4

12. Secondary Outcome: Number of Participants With Maximum Grade 3-5 Toxicities
Description: The maximum grade of toxicities reported by participants over the study duration are tabulated. Per the CTCAE criteria, toxicities are graded on a scale of 0-5, with higher numbers indicating greater severity. The categories correspond as follows:
  3 - severe; 4 - life-threatening; 5 - fatal
Time Frame: 18 months
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants
  0-2 | 34 | 59
  3 | 66 | 47
  4 | 22 | 18
  5 | 10 | 9

13. Secondary Outcome: Infection Type
Description: The number and types of infection events reported are tabulated.
Time Frame: 18 months post-transplant
Population: Infection events
Measure: Count of Units; unit: Infection events
Units Other Than Participants: Infection events
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Number analyzed (Infection events) | 353 | 283
Infection events
  Bacterial | 192 | 161
  Viral | 117 | 95
  Fungal | 37 | 12
  Protozoal | 1 | 0
  Other | 6 | 15

14. Secondary Outcome: Number of Participants With Infections
Description: The maximum severity of infections reported by participants are tabulated.
  The number of infections and the number of patients experiencing infections will be tabulated by type of infection, severity, and time period after transplant. The cumulative incidence of severe, life-threatening, or fatal infections will be compared between the two treatment arms at 6, 12, and 18 months from transplant or until death.
Time Frame: 18 months post-transplant
Population: Transplanted participants
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 132 | 133
Participants
  None | 38 | 43
  Moderate | 42 | 37
  Severe | 40 | 43
  Life Threatening or Fatal | 12 | 10

15. Secondary Outcome: Number of Participants With Cause of Death
Description: Primary cause of death was adjudicated using previously described criteria (Copelan et al. 2007). When relapse occurred, it was considered the primary cause of death regardless of other events.
Time Frame: 18 months post-randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Number analyzed (Participants) | 135 | 137
Participants
  Relapse | 10 | 38
  Organ failure | 3 | 1
  GVHD | 15 | 4
  Infection | 2 | 0
  Sudden death | 0 | 1
  Still alive | 105 | 93

ADVERSE EVENTS:
Time Frame: 18 months post-randomization
Description: Serious Adverse Events (AE) are defined as events associated with death, life-threatening event, disability, congenital anomaly, required intervention to prevent permanent impairment or damage, hospitalization or other serious adverse event. Only unexpected grade 3-5 AEs were required to be reported through the AE system per protocol.
Arm/Group | Myeloablative Conditioning Regimen (MAC) | Reduced Intensity Conditioning (RIC)
Serious Adverse Events (participants affected / at risk) | 21/132 | 16/133
Other Adverse Events (participants affected / at risk) | 7/132 | 4/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Conditioning Regimen (MAC) (N=132) | Reduced Intensity Conditioning (RIC) (N=133)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Immune thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Graft versus host disease (Immune system disorders) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Liver function test increased (Investigations) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 2 (2) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 2 (2) | 0 (0)
Finger amputation (Surgical and medical procedures) | 0 (0) | 1 (1)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 1 (2) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Venoocclusive disease (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Myeloablative Conditioning Regimen (MAC) (N=132) | Reduced Intensity Conditioning (RIC) (N=133)
Chest pain (General disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 2 (2) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Large granular lymphocytosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2014-03-03): https://cdn.clinicaltrials.gov/large-docs/10/NCT01339910/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2015-05-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT01339910/SAP_001.pdf